CLINICAL TRIAL: NCT05602714
Title: Efficacy and Safety of Anterior Cervical Spine Surgery in Patients With Cervical Degenerative Disc Disease - a Real World Data Collection and Analysis Study
Brief Title: Real World Data Collection and Analysis on the Anterior Cervical Spine Surgery
Acronym: ACCSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: KY201402502
Record Dates: First submitted 2022-10-17; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Cervical Disc Degeneration
Keywords: Cervical Degenerative Disease; Cervical Myelopathy; Cervical Radiculopathy; Anterior Cervical Spine Surgery
MeSH Terms: conditions — Radiculopathy | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection Data

SUMMARY:
This observational study aims to evaluate the efficacy and safety of anterior cervical spine surgery in patients with cervical degenerative disc disease

DETAILED DESCRIPTION:
This observational study is an ambispective cohort designed. Patients who are diagnosed cervical degenerative disc disease will be selected to join in this study. Visual Analogue Scale, Japanese Orthopaedic Association Scale, Neck Disability Index, SF-36, and device related or procedure related adverse events will be recorded and compared to evaluate the efficacy and safety of anterior cervical spine surgery in patients with cervical degenerative disc disease

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old
2. Clinical symptoms and imaging support cervical degenerative disc disease；
3. Failed a minimum of 3months conservative treatment
4. Have had (retrospective cohort) or the decision has been made to have (prospective cohort) anterior cervical spine surgery
5. Written informed consent given by subject

Exclusion Criteria:

1. Patients with non-degenerative (e.g., trauma, tumor, and infection) or neuromuscular diseases (e.g., motor neuron disease) were excluded
2. Patients with cervical spine X-ray film and CT scan contraindications
3. Women who are lactating and pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical degenerative disc disease
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Japanese Orthopaedic Association Scale | 1st year
  Establishing criteria for mild, moderate and severe impairment in patients with degenerative cervical myelopathy. The minimum value is 0, and the maximum value is 17. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Neck Disability Index | 1st year
  The index to evaluate the neck pain and life quality. The minimum value is 0%, and the maximum value is 100%. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No